CLINICAL TRIAL: NCT07315698
Title: Efficacy of Oral Paracetamol Compared With Oral Ketoprofen for Pain Management in Office Hysteroscopy: A Double-Blind Randomized Clinical Trial
Brief Title: Efficacy of Oral Paracetamol Compared With Oral Ketoprofen for Pain Management in Office Hysteroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Tricia Dewi Anggraeni, Sp.OG, Subsp. Onk, Associate Professor of Gynecologic Oncology Division, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-08-0983
Record Dates: First submitted 2025-11-14; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2020-10

CONDITIONS: Office Hysteroscopy
Keywords: Office Hysteroscopy; Gynecologic Endoscopy; Outpatient Procedure; Visual Analogue Scale; Non-steroidal Anti-inflammatory Drugs; Women's Health; Analgesic Efficacy
MeSH Terms: interventions — Ketoprofen; Acetaminophen; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketoprofen 100 mg orally for Office Hysteroscopy Pre-Medication (Active Comparator): Ketoprofen 100 mg orally for office hysteroscopy procedure pre-medication 60 minutes before the procedure. Then, assessing the intensity of pain during the procedure and cramping within 30 minutes after the procedure.
  Interventions: Drug: Ketoprofen 100mg
- Paracetamol 1000 mg orally for Office Hysteroscopy Pre-Medication (Active Comparator): Paracetamol 1000 mg orally for office hysteroscopy procedure pre-medication 60 minutes before the procedure. Then, assessing the intensity of pain during the procedure and cramping within 30 minutes after the procedure.
  Interventions: Drug: Paracetamol 1000 Mg Oral Tablet

INTERVENTIONS:
Drug: Ketoprofen 100mg — Ketoprofen 100 mg orally for office hysteroscopy procedure pre-medication 60 minutes before the procedure. Then, assessing the intensity of pain during the procedure and cramping within 30 minutes after the procedure.
  Other Names: Ketoprofen 100mg orally
  Arms: Ketoprofen 100 mg orally for Office Hysteroscopy Pre-Medication
Drug: Paracetamol 1000 Mg Oral Tablet — Paracetamol 1000 mg orally for office hysteroscopy procedure pre-medication 60 minutes before the procedure. Then, assessing the intensity of pain during the procedure and cramping within 30 minutes after the procedure.
  Arms: Paracetamol 1000 mg orally for Office Hysteroscopy Pre-Medication

SUMMARY:
Hysteroscopy is a procedure used to evaluate abnormalities within the uterus (intrauterine. Currently, hysteroscopy can be performed in an outpatient clinic setting according to established standards, known as office hysteroscopy. Although office hysteroscopy offers greater comfort compared with hysteroscopy performed in the operating room, the procedure can still cause pain for patients.

At Dr. Cipto Mangunkusumo National General Hospital, one of the analgesics routinely used for office hysteroscopy is ketoprofen, a non-steroidal anti-inflammatory drug (NSAID) administered rectally. However, ketoprofen frequently causes uncomfortable side effects such as nausea, vomiting, and diarrhea, making alternative analgesics necessary-particularly for patients with contraindications to NSAIDs, including those with allergic reactions. In addition, rectal administration is less practical and less comfortable for patients compared with oral administration.

Therefore, an alternative analgesic with fewer side effects and a more practical route of administration is needed for pain management during office hysteroscopy. Further evaluation is required to assess the efficacy of paracetamol compared with ketoprofen as an alternative analgesic for pain management in office hysteroscopy. Adequate pain management is expected to enhance the overall success of the procedure.

DETAILED DESCRIPTION:
This study will be conducted over a six-months period and involves interview-based data collection and pain assessments integrated with the office hysteroscopy procedure visit. Each participant undergoes an interview of approximately 20 minutes at the beginning of the visit, followed by pain assessments at the time of hysteroscope insertion and again 30 minutes after the procedure is completed.

The study procedures include:

1. Conducting interviews to obtain sociodemographic information, current and past medical history, pregnancy history, medication use, and drug allergy history.
2. Performing a physical examination and additional diagnostic tests to determine the participant's health status.
3. Randomly allocating participants into two groups using simple randomization.
4. Administering analgesic interventions according to group allocation: the first group receives 1000 mg of oral paracetamol, and the second group receives 100 mg of oral ketoprofen, both given one hour before office hysteroscopy. The medications are provided in tablet form and taken with water after a meal.
5. Assessing pain intensity using the Visual Analogue Scale (VAS) at hysteroscope insertion into the external cervical ostium and again 30 minutes after the procedure is completed.
6. Evaluating side effects, patient comfort, and vagal reflexes using validated questionnaires.
7. Recording and analyzing all obtained data.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent an office-hysteroscopy procedure
* Not using analgesics one month before joining the study

Exclusion Criteria:

* Women with a history of Asthma
* Women with a history of Allergy to Paracetamol or NSAID class drugs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
The Intensity of Pain During Office-Hysteroscopy Procedure | During the office-hysteroscopy procedure
  The intensity of pain during office-hysteroscopy procedure, measured using a visual analogue scale when the hysteroscope entered the external cervical ostium

SECONDARY OUTCOMES:
Cramping Pain Score within 30 Minutes After Office-Hysteroscopy Procedure | Within 30 minutes after office-hysteroscopy procedure

CONTACTS AND LOCATIONS:
Locations (1):
- RSCM Kintani, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teran-Alonso MJ, De Santiago J, Usandizaga R, Zapardiel I. Evaluation of pain in office hysteroscopy with prior analgesic medication: a prospective randomized study. Eur J Obstet Gynecol Reprod Biol. 2014 Jul;178:123-7. doi: 10.1016/j.ejogrb.2014.04.030. Epub 2014 May 6. PMID 24835860
- [Background] Hawkey CJ. Non-steroidal anti-inflammatory drugs and peptic ulcers. BMJ. 1990 Feb 3;300(6720):278-84. doi: 10.1136/bmj.300.6720.278. No abstract available. PMID 2106956
- [Background] Tenenbaum J. The epidemiology of nonsteroidal anti-inflammatory drugs. Can J Gastroenterol. 1999 Mar;13(2):119-22. doi: 10.1155/1999/361651. PMID 10203429
- [Background] el Valle, C.; Solano, J.A.; Rodríguez, A.; Alonso, M. Pain management in outpatient hysteroscopy. Gynecol Minim Invasive Ther. 2016;5(4):141-7.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT07315698/Prot_SAP_000.pdf